CLINICAL TRIAL: NCT00210093
Title: A Single-Center, Randomized, Crossover Pharmacokinetic Evaluation of the Effect of Single Doses of Intravenous INS37217, Nasally Inhaled INS37217 and Orally Inhaled INS37217 Solution in Healthy Volunteers
Brief Title: A Pharmacokinetic Evaluation Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 08-106
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
MeSH Terms: interventions — denufosol tetrasodium

INTERVENTIONS:
Drug: denufosol tetrasodium (INS37217)

SUMMARY:
The purpose of this trial is to characterize the pharmacokinetics of INS37217 following intravenous, intranasal, and inhalation administration and to calculate the relative bioavailability of INS37217 when administered via oral or nasal inhalation.

ELIGIBILITY:
Inclusion Criteria:

* Are current nonsmokers or previous smokers who have not smoked within 6 months and who do not have greater than or equal to a 10 pack-year history of tobacco use
* Are within 20% of their ideal body weight
* Are healthy on the basis of a pre-trial physical examination

Exclusion Criteria:

* History or suspicion of recent alcohol, barbiturate, amphetamine or narcotic abuse or a positive urine drug test at study screening
* History of cardiac arrhythmias, any pathological abnormality on the ECG, bronchospasm, diabetes mellitus, thyrotoxicosis, Parkinsonism, asthma, COPD or cardiovascular disease significant drug allergy
* Subject with a physical obstruction in the nose
* Use of concomitant medication other than hormonal contraceptives and multi-vitamins
* Subjects with a current upper respiratory illness or infection for the 2 weeks prior to screening or any chronic respiratory illness

Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-04; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
plasma concentrations of INS37217

SECONDARY OUTCOMES:
Pilot study - not specified

CONTACTS AND LOCATIONS:
Overall Officials: Amy Schaberg, BSN, Study Director